CLINICAL TRIAL: NCT05087797
Title: The Effect of Nicorandil on Left Ventricular Myocardial Strain in Patients With Coronary Chronic Total Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2018253
Record Dates: First submitted 2021-10-10; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nicorandil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nicorandil group (Experimental)
  Interventions: Drug: nicorandil
- control group (No Intervention)

INTERVENTIONS:
Drug: nicorandil — Patients in the nicorandil group were also given nicorandil (Tohoku Nipro Pharmaceutical Corporation, Japan) orally 5 mg three times per day for 3 months
  Arms: nicorandil group

SUMMARY:
Background Nicorandil is recommended as a second-line treatment for stable angina, but randomized-controlled trials (RCTs) to evaluate the benefit of nicorandil for patients with chronic total occlusion (CTO) are still lack.

Objective To determine whether nicorandil can improve left ventricular myocardial strain in patients with CTO.

Methods Patients with CTO were included and were randomized to the nicorandil group and the control group. Nicorandil was given orally 15 mg/day for 3 months in the nicorandil group. 3-dimentional-speckle tracking echocardiography (3D-STE) and the Seattle angina questionnaire (SAQ) survey were performed at baseline and at 3 months. Participants were randomized according to an IBM SPSS23.0-generated randomization schedule, with a 1:1 allocation to the nicorandil group or the control group.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years;1 or more CTO vessels (≥2mm in diameter)

Exclusion Criteria:

* successful PCI for all CTO lesions; ST segment elevation myocardial infarction (STEMI) during the past 3 months; planed coronary artery bypass grafting (CABG) within 3 months; valvular heart disease or congenital heart disease; cardiomyopathy; heart failure with NYHA (New York Heart Association) class III or above; persistent atrial fibrillation or complete left bundle branch block; severe liver, kidney, or lung diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
total area strain | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: ming cui, doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen S, Ma C, Feng X, Cui M. Nicorandil Improves Left Ventricular Myocardial Strain in Patients With Coronary Chronic Total Occlusion. Front Cardiovasc Med. 2022 May 12;9:864223. doi: 10.3389/fcvm.2022.864223. eCollection 2022. PMID 35647043